CLINICAL TRIAL: NCT03569982
Title: Assessing Effectiveness of Acupuncture and Integrative Care in Reducing Anxiety and Pain in Patients Undergoing MOHS Surgery for Dermatological Cancers
Brief Title: Integrative Care and Acupuncture in MOHS Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Clinical associate professor, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CMC-18-0024-CTIL
Record Dates: First submitted 2018-05-02; First posted 2018-06-26 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life
Keywords: Integrative medicine; Peri-operative anxiety; Pain; MOHS surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be referred by the surgeon to MOHS surgery without knowing if integrative care will be provided at the surgery day. Allocation of integrative care to specific surgery days will be determined by a 1:1 randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients receiving best supportive care
- Intervention (Experimental): Patients receiving integrative care (including acupuncture) in addition to best supportive care
  Interventions: Other: Integrative medicine care

INTERVENTIONS:
Other: Integrative medicine care — Including acupuncture, relaxation/breathing, and manual/touch modalities
  Arms: Intervention

SUMMARY:
MOHS method is an effective surgical technique to remove skin cancerous tumors in the head-neck area. Patients undergoing MOHS surgery are struggled with emotional stress during the day of surgery, due to fear of significant damage to the body's image and anxiety about the need for repeated surgeries. In this study we will examine the effect of integrative medicine (including acupuncture, touch/manual, and breathing/relaxation modalities) on the reduction of anxiety and pain in patients undergoing MOHS surgery.

DETAILED DESCRIPTION:
MOHS method is an effective surgical technique to remove skin cancerous tumors in the head-neck area, with immediate microscopic examination in a frozen slice of the full margin. Patients undergoing MOHS surgery are struggled with emotional stress during the day of surgery, due to fear of significant damage to the body's appearance and image and anxiety about the need for repeated surgeries performed on the same day to remove the tumor. In this study we will examine the effect of integrative medicine (including acupuncture, touch/manual, and breathing/relaxation modalities) on the reduction of anxiety and pain in patients undergoing MOHS surgery. The study was designed on the basis of interdisciplinary collaboration of researchers from plastic, integrative and gynecological medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to MOHS surgery

Exclusion Criteria:

* Pregnancy
* Hypertension treated with alpha and beta-blockers
* Chronic atrial fibrillation
* insulin dependent diabetes type 1
* Thyroid disease (hyperthyroidism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Anxiety as assessed by State-Trait Anxiety Inventory | 8 hours
  Alleviating anxiety throughout MOHS surgery

SECONDARY OUTCOMES:
Heart rate variability (HRV) | 30 minutes
  Monitoring HRV
Pain as assessed by visual analogue scale | 60 minutes
  Reducing pain before, during and following local anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided